CLINICAL TRIAL: NCT03439514
Title: A Phase 3, Multinational, Randomized, Placebo-controlled Study of ARRY-371797 (PF-07265803) in Patients With Symptomatic Dilated Cardiomyopathy Due to a Lamin A/C Gene Mutation (REALM-DCM)
Brief Title: A Study of ARRY-371797 (PF-07265803) in Patients With Symptomatic Dilated Cardiomyopathy Due to a Lamin A/C Gene Mutation
Acronym: REALM-DCM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor terminated the study due to futility. The decision to stop the study was not based on safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARRAY-797-301; C4411002 (Other: Alias Study Number); 2017-004310-25 (EudraCT Number)
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Dilated Cardiomyopathy; Lamin A/C Gene Mutation
Keywords: cardiomyopathy; Lamin Type A; heart failure; ARRY-797; C4411002
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Limb-girdle muscular dystrophy, type 1B; Heart Failure | interventions — ARRY-371797

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 parts: a randomized, double-blind treatment period for at least 24 weeks, followed by an ARRY-371797 (PF-07265803) open-label treatment period.
Who Masked: Participant, Investigator
Masking Description: During the randomized, double-blind period, patients, Investigators, site personnel and the sponsor personnel directly involved with the conduct of the study will remain blinded to assigned treatment, except for regulatory reporting requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Double-blind Treatment (Experimental): ARRY-371797 (PF-07265803) tablet orally OR matching placebo tablet orally
  Interventions: Drug: ARRY-371797 (PF-07265803); Other: Placebo
- Part 2 Open-label Treatment (Experimental): ARRY-371797 (PF-07265803) tablet orally
  Interventions: Drug: ARRY-371797 (PF-07265803)

INTERVENTIONS:
Drug: ARRY-371797 (PF-07265803) — 400 mg twice daily (BID)
Other: Placebo — BID
  Arms: Part 1 Double-blind Treatment

SUMMARY:
This is a randomized, double-blind, placebo-controlled study in patients with dilated cardiomyopathy (DCM) due to a mutation of the gene encoding the lamin A/C protein (LMNA). The study will further evaluate a dose level of study drug (ARRY-371797) that has shown preliminary efficacy and safety in this patient population. After the primary analysis has been performed, eligible patients may receive open-label treatment with ARRY-371797.

ELIGIBILITY:
Selected Key Inclusion Criteria:

* Patients with symptomatic lamin A/C protein (LMNA)-related cardiomyopathy Class II/III/ or Class IV defined as:
* Gene positive for a pathogenic, likely pathogenic, or VUS mutation in the LMNA gene as determined by an accredited clinical laboratory.
* Evidence of cardiac impairment in LVEF <= 50%
* Patient will have an implantable cardioverter defibrillator/cardiac resynchronization therapy defibrillator (ICD/CRT-D). ICD implanted at least 4 weeks prior to initiation of study treatment or CRT-D initiated at least 6 months prior to initiation of study treatment and defibrillation function activated at least 4 weeks prior to initiation of study treatment.
* Class II/III patients must have objective functional impairment evidenced by a reduction in 6-minute walk test (6MWT); a. Screening: 6MWT distance >100 m but ≤450 m, AND b. Day -1 visit: 6MWT distance >100 m but ≤485 m, AND c. Baseline visit (Day 1): 6MWT distance >100 m but ≤485
* Class II/III patients must be stable for at least 3 months
* Stable medical and/or device therapy consistent with regional American Heart Association (AHA) / American College of Cardiology (ACC) or European Society of Cardiology (ESC) guidelines at the investigator discretion, without change in heart failure drug(s) dose in the past 1 month.
* Patients must meet acceptable hematology, hepatic and renal laboratory values within 35 days prior to Day 1 as specified in the protocol.

Selected Key Exclusion Criteria:

* Presence of other form(s) of cardiomyopathy contributing to HF (eg, inflammatory or infiltrative cardiomyopathy), clinically significant cardiac anatomic abnormality (eg,LV aneurysm), clinically significant coronary artery disease (eg, coronary revascularization, exercise induced angina) or uncorrected, hemodynamically significant (ie, moderate-severe) primary structural valvular disease not due to HF, per investigator judgment.
* Currently receiving intermittent or continuous IV inotrope infusion, or presence of a ventricular assist device, or history of prior heart transplantation. Participants listed for cardiac transplantation may be enrolled provided transplantation is not likely to occur in the next 6 months.
* Myocardial infarction, cardiac surgical procedures (other than for pacemaker/ICD/CRT-D implantation or replacement), acute coronary syndrome, serious systemic infection with evidence of septicemia, or any major surgical procedure requiring general anesthesia within 3 months prior to screening.
* Currently receiving or deemed at high risk of requiring chronic renal replacement therapy (eg, hemodialysis or peritoneal dialysis) within 6 months.
* Initiation of CRT within 6 months prior to screening.
* Treatment with any investigational agent(s) for HF within 35 days prior to Day 1.
* Malignancy that is active or has been diagnosed within 3 years prior to screening, except surgically curatively resected in situ malignancies or surgically cured early breast cancer, prostate cancer, skin cancer (basal cell carcinoma, squamous cell carcinoma), thyroid cancer, or cervical cancer, or, with prior review by the medical monitor, other early stage surgically curatively resected malignancies with less than a 20% expected 2 year recurrence rate.
* Non-cardiac condition that limits lifespan to < 1 year.
* Serum positive for hepatitis B surface antigen, viremic hepatitis C, or human immunodeficiency virus (HIV) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (106):
- United States (55):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham the Kirklin Clinic, Birmingham, Alabama
  - IDS Pharmacy at UAB Hospital, Birmingham, Alabama
  - Cardiovascular Clinical Trials Unit, Birmingham, Alabama
  - CB Flock Research Corporation, Mobile, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Valley Heart Rhythm Specialists, PLLC, Chandler, Arizona
  - Cardiovascular and Stem Cell Consultants, Gilbert, Arizona
  - Cardiovascular Research Clinic, Gilbert, Arizona
  - Dignity Health, Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Children's Clinic, Tucson, Arizona
  - Banner - Banner University Medical Center South, Tucson, Arizona
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - Banner University Medicine North, Tucson, Arizona
  - Banner University Medical Center Tuscon, Tucson, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Ahmanson Cardiomyopathy Center Cardiovascular Genetics, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Academic Offices Building, Aurora, Colorado
  - University of Colorado Clinical and Translational Research Center, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Innovative Research of West Florida, Clearwater, Florida
  - University of South Florida, Tampa, Florida
  - USF Health, Tampa, Florida
  - Florida Cardiovascular Institute PA, Tampa, Florida
  - Centers for Heart Failure Therapy, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Columbus Cardiology Associates Research - Centricity Research - HyperCore - PPDS, Columbus, Georgia
  - Columbus Cardiology Associates Research - IACT - HyperCore - PPDS, Columbus, Georgia
  - Columbus Regional Research Institute at Talbotton - Centricity Research - HyperCore - PPDS, Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Saint Luke's Idaho Cardiology Associates, Boise, Idaho
  - Brigham and Women's Hospital, Boston, Massachusetts
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Washington University Center For Advanced Medicine, St Louis, Missouri
  - Washington University Center for Outpatient Health, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers New Jersey Medical School - Doctors Office Center, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYU School of Medicine / NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Columbia University/Presbyterian Hospital - Vivian & Seymour Milstein Family Heart Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Stern Cardiovascular Foundation Inc, Germantown, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Baylor Annette C and Harold C Simmons Transplant Institute, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Washington Medical Center, Seattle, Washington
  - Meriter Hospital, Madison, Wisconsin
- Argentina (5):
  - Fundacion Favaloro para la Docencia e Investigacion Medica, Buenos Aires, Buenos Aires F.D.
  - Instituto CAICI, Rosario, Santa Fe Province
  - Hospital Provincial Del Centenario, Rosario, Santa Fe Province
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Hospital Provincial Dr Jose Maria Cullen, Santa Fe
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis, Aalst, Oost-vlaanderen
  - UZ Leuven, Leuven
- Canada (7):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Nova Scotia Health Authority (Capital District Health Authority), Halifax, Nova Scotia
  - NSHA QEII Health Sciences Halifax Infirmary, Halifax, Nova Scotia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Clinical Laboratories of Montreal Heart Institute, Montreal, Quebec
  - Centre Intégré Universitaire de santé et de services sociaux de l'Estrie Centre hospitalier, Sherbrooke, Quebec
- Italy (16):
  - Ospedale Di Cattinara, Trieste, Friuli Venezia Giulia
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Ospedale Santa Maria Della Misericordia Perugia, Perugia - Località S. Andrea Delle Fratte, Perugia
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, PV
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Lacopo Olivotto, Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - A.O.U. di Perugia Ospedale Santa Maria della Misericordia, Perugia, Umbria
  - AO Ospedale Policlinico Consorziale di Bari, Bari
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Pavia - Istituti Clinici Scientifici Maugeri Spa ? Società Benefit, Pavia
  - A.O.U. di Perugia Ospedale Santa Maria Della Misericordia, Perugia
  - A.O.U. di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Presidio Ospedaliero Madonna del Soccorso, San Benedetto del Tronto
  - Ospedale Di Cattinara, Trieste
- Mexico (4):
  - Hospital Boutique Riobamba, Mexico City, Mexico City
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Christus Muguerza Hospital Alta Especialidad, Monterrey, Nuevo León
  - Fundación de Atención e Investigación Médica Lindavista S.C., Mexico City
- Amsterdam UMC, Location Academic Medical Center, Amsterdam, North Holland, Netherlands
- Norway (2):
  - Sykehuset Innlandet HF Hamar, Hamar
  - Oslo University Hospital, Rikshospitalet, Oslo
- Spain (11):
  - Centro de Farmacovigilancia de Galicia, Santiago de Compostela, A Coruña
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario Universitario de Vigo - H. Alvaro Cunqueiro, Vigo, Pontevedra
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital General Universitario Reina Sofia, Córdoba
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Universitario Son Llatzer, Palma de Mallorca
- United Kingdom (3):
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow CITY
  - St Bartholomew's Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Garcia-Pavia P, Lakdawala NK, Sinagra G, Ripoll-Vera T, Afshar K, Priori SG, Ware JS, Owens A, Li H, Angeli FS, Elliott P, MacRae CA, Judge DP. Characterization and natural history of patients with LMNA-related dilated cardiomyopathy in the phase 3 REALM-DCM trial. ESC Heart Fail. 2024 Dec;11(6):4201-4208. doi: 10.1002/ehf2.14955. Epub 2024 Aug 15. PMID 39145700
- [Derived] Garcia-Pavia P, Palomares JFR, Sinagra G, Barriales-Villa R, Lakdawala NK, Gottlieb RL, Goldberg RI, Elliott P, Lee P, Li H, Angeli FS, Judge DP, MacRae CA; REALM-DCM Investigators. REALM-DCM: A Phase 3, Multinational, Randomized, Placebo-Controlled Trial of ARRY-371797 in Patients With Symptomatic LMNA-Related Dilated Cardiomyopathy. Circ Heart Fail. 2024 Jul;17(7):e011548. doi: 10.1161/CIRCHEARTFAILURE.123.011548. Epub 2024 Jul 9. PMID 38979608
- [Derived] Judge DP, Taylor MR, Li H, Oliver C, Angeli FS, Lee PA, MacRae CA. Long-term effectiveness of ARRY-371797 in people with dilated cardiomyopathy and a faulty LMNA gene: a plain language summary. Future Cardiol. 2023 Mar;19(3):117-126. doi: 10.2217/fca-2022-0125. Epub 2023 Apr 3. PMID 37010012
- [Derived] MacRae CA, Taylor MR, Mestroni L, Moses J, Ashley EA, Wheeler MT, Lakdawala NK, Hershberger RE, Sandor V, Saunders ME, Oliver C, Lee PA, Judge DP. Plain Language Summary of Publication of the safety and efficacy of ARRY-371797 in people with dilated cardiomyopathy and a faulty LMNA gene. Future Cardiol. 2023 Feb;19(2):55-63. doi: 10.2217/fca-2022-0099. Epub 2023 Jan 31. PMID 36718638
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-797-301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 77 participants with Lamin A/C protein (LMNA)-related dilated cardiomyopathy (DCM) in New York heart association (NYHA) functional Class II and III were enrolled in the study. All participants enrolled received at least 1 dose of study intervention.
Groups:
- PF-07265803 (ARRY-371797): Participants were randomized to receive PF-07265803 400 mg (4*100 mg tablets) twice daily (BID).
- Placebo: Participants were randomized to receive placebo matched to PF-07265803 BID.
Period: Double-Blind Treatment Period
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Started | 40 | 37
Completed | 0 | 0
Not Completed | 40 | 37
Not completed — Other | 4 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Study Termination by Sponsor | 29 | 32
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 2
Period: Open-Label Treatment Period
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07265803 (ARRY-371797) | Placebo | Total
Number analyzed (Participants) | 40 | 37 | 77
Age, Customized [Count of Participants; unit: Participants]
  18-34 years | 4 | 1 | 5
  35-49 years | 15 | 10 | 25
  50-64 years | 17 | 19 | 36
  >= 65 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 37 | 33 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six-Minute Walk Test (6 MWT) at Week 24
Description: The 6 MWT was an assessment where the distance that a participant could walk on a flat and hard surface in 6 minutes was measured. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed, and under supervision of a qualified professional. Study discontinuation & death were incorporated into endpoint definition through ranking in hypothesis testing of treatment difference. Missing data resulting from study discontinuation were imputed using control-based multiple imputation method to estimate treatment effect.
Time Frame: Baseline, Week 24
Population: Efficacy analysis set (EAS): NYHA functional Class II / III randomized participants. 'Number of Participants Analyzed' = participants evaluable for the outcome measure. Five participants (ARRY-371797 [n=3], placebo [n=2]) discontinued the study before week 24 due to the sponsor's decision to terminate and were excluded from the primary analysis. All participants reported under 'Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row.
Measure: Median (Inter-Quartile Range); unit: Meter
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 37 | 35
Meter
  Baseline: number analyzed (Participants) | 35 | 33
  Baseline | 402.500 [348.195 to 444.000] | 393.935 [360.000 to 425.500]
  Week 24: number analyzed (Participants) | 35 | 33
  Week 24 | 420.234 [358.902 to 459.117] | 393.455 [347.409 to 450.826]
  Week 24 change from baseline: number analyzed (Participants) | 35 | 33
  Week 24 change from baseline | 20.996 [-22.757 to 51.477] | 2.679 [-11.530 to 33.698]
Statistical Analysis 1: Comparison: PF-07265803 (ARRY-371797) vs Placebo; Test type: Superiority; p = 0.818, Van Elteren test — Two-sided p-value; Median Difference (Net) = 4.936, 95% CI 2-sided [-24.246 to 34.118] — The Week 24 change from baseline in 6MWT between PF 07265803 and placebo was estimated using the stratified HL median difference, considering only participants who survived 24 weeks

2. Secondary Outcome: Change From Baseline in 6 MWT at Weeks 4 and 12
Description: The 6 MWT was an assessment where the distance that a participant could walk on a flat and hard surface in 6 minutes was measured. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed, and under supervision of a qualified professional.
Time Frame: Baseline, Week 4, Week 12
Population: EAS included all NYHA functional Class II or III randomized participants. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable for specified rows of respective arms.
Measure: Median (Full Range); unit: Meter
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Meter
  Change at Week 4: number analyzed (Participants) | 35 | 32
  Change at Week 4 | 15.40 [-72.0 to 71.8] | -2.60 [-85.0 to 34.5]
  Change at Week 12: number analyzed (Participants) | 33 | 33
  Change at Week 12 | 21.47 [-70.2 to 69.3] | 10.00 [-100.9 to 89.5]

3. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Physical Limitation (PL) and Total Symptom Score (TSS) Domain Scores at Weeks 12 and 24
Description: The KCCQ measured the effects of symptoms, functional (physical) limitations, and psychological distress on an individual's health-related quality of life. It contains 23 items, which assessed the ability to perform activities of daily living, frequency and severity of symptoms, the impact of these symptoms, and health-related quality of life. PL was a single questionnaire with score range of 0 to 100, where higher scores reflected better physical functioning status. TSS included frequency and severity of symptoms, and the impact of these symptoms. TSS scores were transformed to a range of 0 to 100, where higher scores reflected better health status.
Time Frame: Baseline, Week 12, Week 24
Population: EAS included all NYHA functional Class II or III randomized participants. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Units on a scale
  Week 12 Physical Limitation (PL): number analyzed (Participants) | 33 | 32
  Week 12 Physical Limitation (PL) | 4.48 (11.373) | -1.17 (15.326)
  Week 24 Physical Limitation (PL): number analyzed (Participants) | 28 | 31
  Week 24 Physical Limitation (PL) | 2.98 (17.510) | 1.21 (14.104)
  Week 12 Total Symptom Score (TSS): number analyzed (Participants) | 33 | 32
  Week 12 Total Symptom Score (TSS) | 3.66 (12.487) | 1.04 (16.491)
  Week 24 Total Symptom Score (TSS): number analyzed (Participants) | 28 | 31
  Week 24 Total Symptom Score (TSS) | 4.02 (19.171) | -0.94 (14.981)

4. Secondary Outcome: Number of Participants With Improvement From Baseline in Patient Global Impression of Severity (PGI-S) Score at Weeks 12 and 24
Description: PGI-S is a global index that rate the severity of the disease using a 5-point scale. In this outcome the number of participants with improvements in PGI-S the severity of their heart failure symptoms and in the severity of their PL were reported. Measured by the scale of: none, mild, moderate, severe or very severe (listed from better to worse).
Time Frame: Week 12, Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Week 12: Severity of heart failure symptoms: number analyzed (Participants) | 33 | 32
  Week 12: Severity of heart failure symptoms: None | 4 | 5
  Week 12: Severity of heart failure symptoms: Mild | 16 | 14
  Week 12: Severity of heart failure symptoms: Moderate | 8 | 10
  Week 12: Severity of heart failure symptoms: Severe | 4 | 2
  Week 12: Severity of heart failure symptoms: Very Severe | 1 | 1
  Week 24: Severity of heart failure symptoms: number analyzed (Participants) | 28 | 31
  Week 24: Severity of heart failure symptoms: None | 4 | 6
  Week 24: Severity of heart failure symptoms: Mild | 11 | 10
  Week 24: Severity of heart failure symptoms: Moderate | 10 | 12
  Week 24: Severity of heart failure symptoms: Severe | 3 | 3
  Week 24: Severity of heart failure symptoms: Very Severe | 0 | 0
  Week 12: Severity of physical activity limitations: number analyzed (Participants) | 33 | 32
  Week 12: Severity of physical activity limitations: None | 6 | 7
  Week 12: Severity of physical activity limitations: Mild | 11 | 5
  Week 12: Severity of physical activity limitations: Moderate | 12 | 15
  Week 12: Severity of physical activity limitations: Severe | 3 | 4
  Week 12: Severity of physical activity limitations: Very Severe | 1 | 1
  Week 24: Severity of physical activity limitations: number analyzed (Participants) | 28 | 31
  Week 24: Severity of physical activity limitations: None | 6 | 6
  Week 24: Severity of physical activity limitations: Mild | 5 | 7
  Week 24: Severity of physical activity limitations: Moderate | 13 | 15
  Week 24: Severity of physical activity limitations: Severe | 4 | 3
  Week 24: Severity of physical activity limitations: Very Severe | 0 | 0

5. Secondary Outcome: Number of Participants With Improvement From Baseline in Patient Global Impression of Change (PGI-C) Score at Weeks 12 and 24
Description: PGI-C is a global index that rate the severity of the disease using a 7-point scale. In this outcome the number participants with improvements in their heart failure symptoms and "in their physical activity limitations?", were reported. Measured by the scale of: very much better, moderately better, a little better, no change, a little worse, moderately worse, very much worse (listed from better to worse).
Time Frame: Week 12, Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Week 12: Overall change in heart failure symptoms: number analyzed (Participants) | 33 | 32
  Week 12: Overall change in heart failure symptoms: Very Much Better | 0 | 2
  Week 12: Overall change in heart failure symptoms: Moderately Better | 3 | 1
  Week 12: Overall change in heart failure symptoms: A Little Better | 7 | 9
  Week 12: Overall change in heart failure symptoms: No Change | 18 | 17
  Week 12: Overall change in heart failure symptoms: A Little Worse | 3 | 1
  Week 12: Overall change in heart failure symptoms: Moderately Worse | 1 | 0
  Week 12: Overall change in heart failure symptoms: Very Much Worse | 1 | 2
  Week 24: Overall change in heart failure symptoms: number analyzed (Participants) | 28 | 29
  Week 24: Overall change in heart failure symptoms: Very Much Better | 1 | 1
  Week 24: Overall change in heart failure symptoms: Moderately Better | 3 | 2
  Week 24: Overall change in heart failure symptoms: A Little Better | 7 | 6
  Week 24: Overall change in heart failure symptoms: No Change | 16 | 16
  Week 24: Overall change in heart failure symptoms: A Little Worse | 0 | 2
  Week 24: Overall change in heart failure symptoms: Moderately Worse | 1 | 1
  Week 24: Overall change in heart failure symptoms: Very Much Worse | 0 | 1
  Week 12: Overall change in physical activity limitations: number analyzed (Participants) | 33 | 32
  Week 12: Overall change in physical activity limitations: Very Much Better | 0 | 1
  Week 12: Overall change in physical activity limitations: Moderately Better | 3 | 2
  Week 12: Overall change in physical activity limitations: A Little Better | 3 | 5
  Week 12: Overall change in physical activity limitations: No Change | 24 | 21
  Week 12: Overall change in physical activity limitations: A Little Worse | 0 | 1
  Week 12: Overall change in physical activity limitations: Moderately Worse | 3 | 1
  Week 12: Overall change in physical activity limitations: Very Much Worse | 0 | 1
  Week 24: Overall change in physical activity limitations: number analyzed (Participants) | 28 | 29
  Week 24: Overall change in physical activity limitations: Very Much Better | 1 | 1
  Week 24: Overall change in physical activity limitations: Moderately Better | 3 | 0
  Week 24: Overall change in physical activity limitations: A Little Better | 3 | 4
  Week 24: Overall change in physical activity limitations: No Change | 19 | 20
  Week 24: Overall change in physical activity limitations: A Little Worse | 1 | 3
  Week 24: Overall change in physical activity limitations: Moderately Worse | 1 | 1
  Week 24: Overall change in physical activity limitations: Very Much Worse | 0 | 0

6. Secondary Outcome: Change From Baseline in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) at Weeks 4, 12, and 24
Description: NT pro-BNP is a cardiac biomarker that is released in the blood in response to changes in the pressure inside of the heart. Levels go up when heart failure develops or gets worse, and levels go down when heart failure is stable or improves. This biomarker helps to measure the changes in the severity of heart failure over time in response to therapy.
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomoles per liter
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
picomoles per liter
  Change at Week 4: number analyzed (Participants) | 33 | 33
  Change at Week 4 | -43.89 (65.465) | -3.07 (62.745)
  Change at Week 12: number analyzed (Participants) | 31 | 32
  Change at Week 12 | -36.40 (69.228) | -0.70 (54.870)
  Change at Week 24: number analyzed (Participants) | 23 | 28
  Change at Week 24 | 5.00 (236.643) | 24.37 (134.225)

7. Secondary Outcome: Composite Time to First Occurrence of All-Cause Mortality or Worsening Heart Failure (WHF)
Description: Defined as the time from randomization to the first occurrence of any event of death due to any cause, or worsening heart failure (HF-related hospitalization or HF-related urgent care visit). Kaplan-Meier method and cox regression model were used for analysis.
Time Frame: Maximum up to 212.28 weeks (maximum exposure was 208 weeks)
Population: The safety analysis set (SAS) included all participants who received at least 1 dose of study intervention regardless of NYHA functional class.
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Events
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Number analyzed (Events) | 3 | 7
Weeks | NA [NA to NA] — Median and 95% CI could not be estimated as there were very few participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated as there were very few participants with events.
Statistical Analysis 1: Comparison: PF-07265803 (ARRY-371797) vs Placebo; Test type: Other; p = 0.2257, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.13 to 1.39]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from randomization to death due to any cause. Participants who did not have a death date were censored for OS at their last contact date. Kaplan-Meier method and cox regression model were used for analysis.
Time Frame: From randomization up to death due to any cause or censored date, maximum up to 212.28 weeks (maximum exposure was of 208 weeks)
Population: The SAS included all participants who received at least 1 dose of study intervention regardless of NYHA functional class.
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Events
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Number analyzed (Events) | 3 | 3
Weeks | NA [NA to NA] — Median and 95% CI could not be estimated as there were very few participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated as there were very few participants with events.
Statistical Analysis 1: Comparison: PF-07265803 (ARRY-371797) vs Placebo; Test type: Other; p = 0.8370, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.30 to 4.63]

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and by Severity
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and all Non-SAEs. Grade >=3 AEs meant severe AEs.
Time Frame: Maximum up to 212.28 weeks (maximum exposure was of 208 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Participants with TEAEs | 35 | 34
  Participants with serious TEAEs | 10 | 21
  Participants with severe (Grades >=3) TEAEs | 16 | 20

10. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (eosinophils, erythrocytes, hemoglobin, hematocrit, granulocytes, leukocytes, lymphocytes, monocytes, platelets, neutrophils, nucleated erythrocytes); blood chemistry (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, C-reactive protein, calcium, chloride, creatinine, creatine kinase, epidermal growth factor receptor, follicle stimulating hormone, gamma glutamyl transferase, glucose, magnesium, N-Terminal ProB-type natriuretic peptide, phosphate, potassium, protein, sodium, potassium, thyrotropin, troponin I, troponin T, urate).
Time Frame: Maximum up to 212.28 weeks (maximum exposure was of 208 weeks)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Eosinophils: High (>0.8) 10^9/L | 1 | 0
  Eosinophils/Leukocytes: High (>7) % | 1 | 1
  Erythrocyte Mean Corpuscular Hemoglobin Concentration: Low (<310) g/L | 30 | 29
  Erythrocyte Mean Corpuscular Hemoglobin: Low (<27) pg | 6 | 3
  Erythrocyte Mean Corpuscular Hemoglobin: High (>34) pg | 0 | 1
  Erythrocyte Mean Corpuscular Volume: Low (Males <78, Females <82) | 2 | 2
  Erythrocyte Mean Corpuscular Volume: High (Males >100, Females >102) | 10 | 15
  Erythrocytes: Low (Males: < 4.63, Females: <3.7) 10^12/L | 14 | 16
  Erythrocytes: High (Males: > 6.08, Females: > 5.2) 10^12/L | 4 | 4
  Erythrocytes Distribution Width: High (>14.5) % | 22 | 20
  Hematocrit: Low (Males: <0.37, Females: <0.33) L/L | 1 | 3
  Hematocrit: High (Males: >0.51, Females: >0.47) L/L | 12 | 15
  Hemoglobin: Low (Males: < 125; Females: <110) g/L | 7 | 5
  Hemoglobin: High (Males: > 170; Females: > 155) g/L | 5 | 4
  Immature Granulocytes: High (> 0.07) 10^9/L | 9 | 7
  Immature Granulocytes/Leukocytes: High (> 1) % | 6 | 6
  Leukocytes: Low (< 3.7) 10^9/L | 1 | 0
  Leukocytes: High (> 11) 10^9/L | 9 | 8
  Lymphocytes: Low (< 0.9) 10^9/L | 3 | 4
  Lymphocytes: Low (> 3.6) 10^9/L | 4 | 2
  Lymphocytes/Leukocytes: Low (< 12) % | 3 | 3
  Lymphocytes/Leukocytes: High (> 46) % | 2 | 1
  Mean Platelet Volume: Low (< 9.6) fL | 5 | 0
  Mean Platelet Volume: High (> 13.8) fL | 3 | 3
  Monocytes: High (> 1.2) 10^9/L | 1 | 1
  Monocytes/Leukocytes: High (>11) % | 11 | 10
  Neutrophils: LOW (< 1.7) 10^9/L | 1 | 1
  Neutrophils: HIGH (> 7.9) 10^9/L | 8 | 5
  Neutrophils/Leukocytes: HIGH (> 71) % | 16 | 17
  Nucleated Erythrocytes: HIGH (> 0.01) 10^9/L | 6 | 1
  Nucleated Erythrocytes/Leukocytes: HIGH (> 0.2) % | 6 | 1
  Platelets: LOW (< 163) 10^9/L | 13 | 11
  Platelets: HIGH (> 375) 10^9/L | 2 | 1
  Alanine Aminotransferase: LOW (< 10) U/L | 4 | 5
  Alanine Aminotransferase: HIGH (Males: > 40; Females: > 33) U/L | 18 | 17
  Albumin: LOW (< 35) g/L | 1 | 0
  Alkaline Phosphatase: LOW (Males: < 43; Females: <30) U/L | 3 | 5
  Alkaline Phosphatase: HIGH (> 115) U/L | 4 | 5
  Aspartate Aminotransferase: HIGH (Males: > 43; Females: > 36) U/L | 11 | 8
  Bicarbonate: LOW (< 21) mmol/L | 9 | 12
  Bicarbonate: HIGH (> 33) mmol/L | 0 | 1
  Bilirubin: HIGH (> 18.8) mcmol/L | 4 | 12
  Blood Urea Nitrogen: HIGH (> 7.14) mmol/L | 28 | 27
  C Reactive Protein: HIGH (> 47.6) nmol/L | 20 | 19
  Calcium: LOW (< 2.12) mmol/L | 0 | 1
  Calcium: HIGH (> 2.62) mmol/L | 0 | 1
  Chloride: LOW (< 95) mmol/L | 2 | 1
  Creatine Kinase: LOW (< 24) U/L | 0 | 2
  Creatine Kinase: HIGH (Males: > 207; Females: > 169) U/L | 20 | 12
  Creatinine: LOW (< 62) mcmol/L | 14 | 13
  Creatinine: HIGH (> 124) mcmol/L | 4 | 6
  Creatinine Clearance: LOW (Males: < 85; Females: <75) mL/min | 9 | 8
  Creatinine Clearance: HIGH (Males: > 125; Females: > 115) mL/min | 16 | 14
  Direct Bilirubin: HIGH (> 6.8) mcmol/L | 4 | 8
  Epidermal Growth Factor Receptor: LOW (Males: < 60) mL/min/1.73m2 | 1 | 0
  Follicle Stimulating Hormone: HIGH (Males: > 12.4; Females: > 21.5) IU/L | 2 | 4
  Gamma Glutamyl Transferase: LOW (Males: < 10; Females: <5) U/L | 1 | 0
  Gamma Glutamyl Transferase: HIGH (Males: > 49; Females: > 32) U/L | 15 | 27
  Glucose: LOW (Males < 3.94, Females < 3.33) mmol/L | 4 | 4
  Glucose: HIGH (Males > 7.66, Females > 6.38) mmol/L | 10 | 10
  Magnesium: HIGH (> 1.05) mmol/L | 1 | 1
  N-Terminal ProB-type Natriuretic Peptide: HIGH (> 14.63) pmol/L | 40 | 37
  Phosphate: LOW (< 0.81) mmol/L | 6 | 6
  Phosphate: HIGH (> 1.45) mmol/L | 8 | 4
  Potassium: LOW (< 3.5) mmol/L | 1 | 0
  Potassium: HIGH (> 5) mmol/L | 7 | 16
  Protein: LOW (< 60) g/L | 2 | 3
  Protein: High (> 80) g/L | 2 | 3
  Sodium: HIGH (> 145) mmol/L | 1 | 1
  Thyrotropin: LOW (< 0.27) mIU/L | 1 | 1
  Thyrotropin: HIGH (> 4.2) mIU/L | 5 | 5
  Troponin I: HIGH (> 0.3) mcg/L | 4 | 6
  Troponin T: HIGH (> 14) ng/L | 36 | 34
  Urate: LOW (Males: < 0.238; Females: <0.119) mmol/L | 3 | 2
  Urate: HIGH (Males: > 0.476; Females: > 0.357) mmol/L | 9 | 17

11. Secondary Outcome: Number of Participants According to Categorization of Abnormal Vital Signs
Description: Following vital sign parameters were assessed: diastolic blood pressure, systolic blood pressure, heart rate, and body weight. Vital sign abnormalities criteria included: a) systolic blood pressure (mmHg): decrease (change <= -20, or value <90) and increase (change >=20, or value >140); b) diastolic blood pressure (mmHg): decrease (change <= -15, or value <60) and increase (change >=15, or value >90); c) heart Rate (bpm) decrease: (change <= -15, or value <50) and increase (change >=15, or value >100); d) weight: (kg) decrease (Change <= -7%) and increase (Change > =7%).
Time Frame: Maximum up to 212.28 weeks (maximum exposure was of 208 weeks)
Population: The SAS included all participants who received at least 1 dose of study intervention regardless of NYHA functional class. Here, "Number Analyzed" signifies number of participants evaluable for specified rows of respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Systolic Blood Pressure (mmHg): Decrease: number analyzed (Participants) | 37 | 37
  Systolic Blood Pressure (mmHg): Decrease | 22 | 17
  Systolic Blood Pressure (mmHg): Increase: number analyzed (Participants) | 37 | 37
  Systolic Blood Pressure (mmHg): Increase | 6 | 14
  Diastolic Blood Pressure (mmHg): Decrease: number analyzed (Participants) | 37 | 37
  Diastolic Blood Pressure (mmHg): Decrease | 28 | 22
  Diastolic Blood Pressure (mmHg): Increase: number analyzed (Participants) | 37 | 37
  Diastolic Blood Pressure (mmHg): Increase | 7 | 18
  Heart Rate (bpm): Decrease: number analyzed (Participants) | 37 | 37
  Heart Rate (bpm): Decrease | 7 | 9
  Heart Rate (bpm): Increase: number analyzed (Participants) | 37 | 37
  Heart Rate (bpm): Increase | 15 | 10
  Weight (kg): Decrease: number analyzed (Participants) | 36 | 35
  Weight (kg): Decrease | 10 | 7
  Weight (kg): Increase: number analyzed (Participants) | 36 | 35
  Weight (kg): Increase | 5 | 1

12. Secondary Outcome: Number of Participants According to Categorization of Electrocardiogram (ECG) Data
Description: Following parameters were analyzed: heart rate, QT interval, corrected QT (QTc) interval, Bazett's correction QT (QTcB) interval, and Fridericia's correction (QTcF) interval. Criteria for notable ECG values were as follows: QT interval (in millisecond [msec]) new (newly occurring post-baseline value) greater than (>) 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Fredericia formula (QTcF) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Bazett's formula (QTcB) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; heart rate in bpm new (newly occurring post-baseline value) <60 and >100.
Time Frame: Maximum up to 212.28 weeks (maximum exposure was of 208 weeks)
Population: The SAS included all participants who received at least 1 dose of study intervention regardless of NYHA functional class. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows of respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 28 | 26
Participants
  QTcB (msec): New >450: number analyzed (Participants) | 10 | 6
  QTcB (msec): New >450 | 5 | 4
  QTcB (msec): New >480: number analyzed (Participants) | 17 | 15
  QTcB (msec): New >480 | 10 | 4
  QTcB (msec): New >500: number analyzed (Participants) | 23 | 18
  QTcB (msec): New >500 | 11 | 2
  QTcB (msec): Increase from baseline >30 | 12 | 4
  QTcB (msec): Increase from baseline >60 | 5 | 1
  QTcF (msec): New >450: number analyzed (Participants) | 10 | 6
  QTcF (msec): New >450 | 7 | 2
  QTcF (msec): New >480: number analyzed (Participants) | 18 | 17
  QTcF (msec): New >480 | 9 | 3
  QTcF (msec): New >500: number analyzed (Participants) | 24 | 20
  QTcF (msec): New >500 | 8 | 4
  QTcF (msec): Increase from baseline >30 | 11 | 4
  QTcF (msec): Increase from baseline >60 | 3 | 0
  QT (msec): New >450: number analyzed (Participants) | 9 | 10
  QT (msec): New >450 | 5 | 4
  QT (msec): New >480: number analyzed (Participants) | 21 | 18
  QT (msec): New >480 | 11 | 1
  QT (msec): New >500: number analyzed (Participants) | 24 | 22
  QT (msec): New >500 | 2 | 1
  QT (msec): Increase from baseline >30 | 8 | 3
  QT (msec): Increase from baseline >60 | 2 | 0
  Heart rate (bpm): New <60: number analyzed (Participants) | 18 | 19
  Heart rate (bpm): New <60 | 1 | 0

13. Secondary Outcome: Number of Participants With a New Clinically Significant Ventricular or Atrial Arrhythmias
Description: Arrhythmia assessment: incidence of new and clinically significant ventricular or atrial arrhythmias was assessed by an implantable cardioverter defibrillator (ICD) or CRT defibrillator (CRT-D) applicable device interrogations.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
Number analyzed (Participants) | 40 | 37
Participants
  Baseline: Clinically significant atrial arrhythmia: number analyzed (Participants) | 29 | 25
  Baseline: Clinically significant atrial arrhythmia | 0 | 0
  Week 12: Clinically significant atrial arrhythmia: number analyzed (Participants) | 20 | 20
  Week 12: Clinically significant atrial arrhythmia | 0 | 2
  Week 24: Clinically significant atrial arrhythmia: number analyzed (Participants) | 14 | 15
  Week 24: Clinically significant atrial arrhythmia | 0 | 0
  Baseline: Clinically significant ventricular arrhythmia: number analyzed (Participants) | 24 | 24
  Baseline: Clinically significant ventricular arrhythmia | 0 | 0
  Week 12: Clinically significant ventricular arrhythmia: number analyzed (Participants) | 18 | 18
  Week 12: Clinically significant ventricular arrhythmia | 0 | 3
  Week 24: Clinically significant ventricular arrhythmia: number analyzed (Participants) | 14 | 15
  Week 24: Clinically significant ventricular arrhythmia | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day1) up to a maximum of 208 weeks
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. All participants who receive any of the study intervention.
Arm/Group | PF-07265803 (ARRY-371797) | Placebo
All-Cause Mortality (participants affected / at risk) | 3/40 | 3/37
Serious Adverse Events (participants affected / at risk) | 10/40 | 21/37
Other Adverse Events (participants affected / at risk) | 31/40 | 27/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-07265803 (ARRY-371797) (N=40) | Placebo (N=37)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (3) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 5 (8) | 5 (6)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-07265803 (ARRY-371797) (N=40) | Placebo (N=37)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 5 (10)
Atrial flutter (Cardiac disorders) | 3 (4) | 2 (5)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 7 (10) | 8 (12)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (6)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 12 (19) | 4 (7)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (7)
Stomatitis (Gastrointestinal disorders) | 5 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 3 (4)
Fatigue (General disorders) | 4 (5) | 3 (6)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 11 (14) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 9 (13) | 4 (4)
Headache (Nervous system disorders) | 4 (6) | 6 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (8)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT03439514/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03439514/SAP_001.pdf